CLINICAL TRIAL: NCT00344201
Title: Assessment of Fibrin Glue in Pterygium Surgery and Other Forms of Ocular Surface Reconstruction
Brief Title: Assessment of Fibrin Glue in Pterygium Surgery and Other Forms of External Eye Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National University of Singapore (Other)
Responsible Party: Yong Ming Por, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R389/47/2004
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Pterygium; Ocular Surface Cicatrizing Diseases
Keywords: Pterygium; Fibrin adhesive; Conjunctival graft; Ocular surface reconstruction
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Tisseel fibrin adhesive — Intraoperative application to scleral bed and graft

SUMMARY:
Tisseel fibrin adhesive has been used extensively in many forms of surgery. Its use in eye surgery has been relatively recent. A few studies recently showed it was effective in securing conjunctival grafts in pterygium surgery, and in securing wounds after glaucoma and squint surgery.

We sought to confirm its effectiveness in pterygium surgery, as well as prove its effectiveness in securing other material to the ocular surface such as amniotic membrane. Our hypothesis is that fibrin adhesive is effective in securing various types of material to the ocular surface for a sufficient length of time to allow adequate healing before it is absorbed and degraded.

DETAILED DESCRIPTION:
AIMS OF STUDY:

This project seeks to evaluate the efficacy of fibrin glue (Tisseel) as an alternative to conventional sutures in ocular surface reconstruction, including pterygium excision with conjunctival autografting and other forms of conjunctival and amniotic membrane surgery.

It aims to evaluate the safety and efficacy of fibrin glue in pterygium and other forms of ocular surface conjunctival and amniotic membrane surgery, as an alternative to conventional suturing. We will perform conjunctival autografting in 30 patients with primary or recurrent pterygium, and in addition, up to 20 patients undergoing either conjunctival or amniotic membrane ocular surface reconstruction for a variety of diverse ocular surface disorders including persistent epithelial defects, Stevens Johnson syndrome, chemical and thermal burns and other fornix shortening/symblepharon conditions. Efficacy endpoints will be the ability of fibrin glue to form stable adherence of the conjunctival/AM graft postoperatively, and in cases of pterygium, the percentage of pterygium recurrence at 6 months following surgery, and subjective indications of postoperative comfort/discomfort. Safety data will include the close monitoring of any potential side-effects including graft loss, infection, pain/discomfort, excessive ocular surface inflammation, epithelial breakdown, and any complications resulting in visual loss. Patients will not be charged for the fibrin glue.

If successful, the use of fibrin glue will be a useful adjunct in ocular surface reconstruction, reducing time of surgery and suture-related complications and discomfort. The cost-benefit ratio will need to be examined, but full-paying patients who can afford it may be offered fibrin glue in pterygium surgery as a surgical option.

Study Plan

This will be a non-randomized prospective series of surgical cases of pterygium surgery or ocular surface reconstruction in which the viability and efficacy of fibrin glue in replacing or augmenting sutures will be evaluated.

Patient Numbers and Selection

1. Pterygium cases: Patients will be referred by SNEC doctors to the Corneal Clinic for study counseling and enrolment. Up to 30 cases of either primary or recurrent pterygium requiring pterygium excision with conjunctival autografting will be counseled for study inclusion. The potential benefits and risks of using fibrin glue as opposed to conventional sutures will be explained with full informed consent. All surgery will be performed by the PI.
2. Other ocular surface reconstructions: Up to 20 cases of ocular surface reconstruction from the SNEC Corneal Clinic requiring suturing of conjunctival grafts or AM will be counseled for study inclusion. Significant variations in diagnosis and indications exist for ocular surface transplantation and are too numerous to elucidate, but cases will generally include ocular surface and fornix reconstructions following symblepharon and cicatrizing disorders, chemical and thermal burns, etc. The potential benefits and risks of using fibrin glue as opposed to conventional sutures will be explained with full informed consent. All surgery will be performed by the PI.

All patients will be followed up at 1 day post-operatively, 1 week, 1 month, 3 months and 6 months. Regular slit-lamp anterior segment photography and detailed recording of the status of the grafts will be performed.

Procedures and Data Collection

The patients will be fully informed of the aim and procedures of the study.

The following data will be captured:

1. Visual acuity on standard Snellen chart
2. Pterygium Grading (T1-3)
3. Documentation of pterygium location, primary or recurrent status
4. Slit-lamp photography, pre- and post-surgery
5. subjective assessment of postoperative discomfort
6. Practical benefits anticipated from successfully completed project (1/2 page)

If successful, the use of fibrin glue will be a useful adjunct in ocular surface reconstruction, significantly reducing surgical time, and obviating suture-related complications and discomfort. The cost-benefit ratio will need to be examined, but full-paying patients who can afford it may be offered fibrin glue in pterygium surgery as a surgical option. Up to 3 consecutive cases can be performed with one Tisseel unit.

ELIGIBILITY:
Inclusion Criteria:

1. significant pterygium clinically requiring excision
2. willingness to participate in research project and to attend research clinic

Exclusion Criteria:

1. age < 18 years
2. other concurrent corneal pathology
3. poor acuity due to other ocular pathology
4. poor general health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-11; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Graft dislocation | 3 months
Pterygium recurrence | 6 months

SECONDARY OUTCOMES:
Graft dimensions | 6 months
Patient comfort on visual analogue scale | 1 month
Visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald TH Tan, FRCOphth, Principal Investigator — Singapore Eye Research Institute; Yong M Por, FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Background] Tan DT, Chee SP, Dear KB, Lim AS. Effect of pterygium morphology on pterygium recurrence in a controlled trial comparing conjunctival autografting with bare sclera excision. Arch Ophthalmol. 1997 Oct;115(10):1235-40. doi: 10.1001/archopht.1997.01100160405001. PMID 9338666
- [Background] Koranyi G, Seregard S, Kopp ED. Cut and paste: a no suture, small incision approach to pterygium surgery. Br J Ophthalmol. 2004 Jul;88(7):911-4. doi: 10.1136/bjo.2003.032854. PMID 15205236
- [Background] Cohen RA, McDonald MB. Fixation of conjunctival autografts with an organic tissue adhesive. Arch Ophthalmol. 1993 Sep;111(9):1167-8. doi: 10.1001/archopht.1993.01090090017006. No abstract available. PMID 8363455
- [Background] Biedner B, Rosenthal G. Conjunctival closure in strabismus surgery: Vicryl versus fibrin glue. Ophthalmic Surg Lasers. 1996 Nov;27(11):967. PMID 8938809
- [Background] Schlag G , Redl H. Fibrin Sealant in Operative Medicine. Vol 2.Ophthalmology, neurosurgery. Berlin, Heidelberg: Springer Verlag, 1986.